CLINICAL TRIAL: NCT06536231
Title: Hemodynamic Variations During Remote Ischemic Conditioning in Critical Ill Patients
Acronym: HERICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Andrius Pranskunas, prof., Lithuanian University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1.2
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Critical Illness
Keywords: Remote ischemic conditioning; Passive leg raising; Hemodynamic; Perfusion index; Fluid responsiveness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Passive leg raising and Remote ischemic conditioning (Experimental): Supine position was followed by the passive leg raising (PLR) maneuver. After completing the PLR test, participants were placed in the supine position for 5 min. Thereafter, remote ischemic conditioning (RIC) was performed. After the RIC procedure, the patient is left in supine position for 5 minutes. Then the PLR test was repeated, after which the participants were placed in a supine position for another 5 min at rest. When the patient fluid responder, physician in charge may decide to perform a fluid infusion (500 mL of crystaloids). The PLR test can also be performed to make decision for fluid removal. This decision is triggered by a negative PLR test in the later phase of ICU treatment. If the physician has decided to administer a fluids, systemic hemodynamics and peripheral perfusion index are measured immediately after completion of the fluid infusion.
  Interventions: Procedure: Remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) procedure comprise three repetitions of brachial cuff inflation to 200 mmHg for five minutes following deflation to 0 mmHg for another five minutes. The procedure overall took 30 minutes.

SUMMARY:
The main objectives of this study are to evaluate the changes in hemodynamics occurring during the remote ischemic conditioning (RIC) procedure and to compare the hemodynamic responses elicited by passive leg raising before and after the RIC intervention.

DETAILED DESCRIPTION:
The investigators hypothesized that the inflation of the blood pressure cuff during the remote ischemic conditioning (RIC) procedure would lead to an increase in stroke volume (SV), cardiac index (CI), and peripheral perfusion index and that these changes would correlate with the hemodynamic changes induced by passive leg raising (PLR).

Furthermore, the clinical relevance of the RIC effect in critically ill patients, particularly in terms of determining their hemodynamic responsiveness, remains uncertain. The investigators hypothesized that the RIC procedure influences hemodynamic changes during PLR.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years,
* admitted to the intensive care unit,
* monitored with a transpulmonary thermodilution device with calibrated pulse contour analysis (Pulsion Medical Systems, Munich, Germany),
* decision by the physician in charge to perform passive leg raising.

Exclusion Criteria:

* pregnancy,
* advanced malignancy,
* peripheral artery disease affecting both arms,
* head trauma,
* deep vein thrombosis in the lower limbs,
* intra-abdominal hypertension, defined as an intra-abdominal pressure greater than 12 mmHg.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximal change in stroke volume index during remote ischemic conditioning (RIC) procedure | During RIC procedure
  Change in this parameter is determined during each inflation and release of the blood pressure cuff.
Maximal change in cardiac index during RIC procedure | During RIC procedure
  Change in this parameter is determined during each inflation and release of the blood pressure cuff.
Maximal change in peripheral perfusion index during RIC procedure | During RIC procedure
  Change in this parameter is determined during each inflation and release of the blood pressure cuff. The perfusion index is measured on a hand that is not equipped with a blood pressure cuff.
The correlation between the maximal changes in stroke volume index, cardiac index, and peripheral perfusion index observed during the RIC procedure and those observed during passive leg raising (PLR). | During RIC procedure, as well as during passive leg raising.
  The maximum changes in these parameters, as determined by the RIC procedure and PLR, were identified, and their correlation was subsequently calculated. The perfusion index is measured on a hand that is not equipped with a blood pressure cuff.
The correlation between the maximal changes in stroke volume index, cardiac index, and peripheral perfusion index observed during PLR before the RIC procedure and those observed during PLR after the RIC procedure. | During PLR both before and after the RIC procedure.
  The maximum changes in these parameters, as measured during PLR before and after the RIC procedure, were identified. Subsequently, the correlation between these changes was calculated. The perfusion index is measured on a hand that is not equipped with a blood pressure cuff.

SECONDARY OUTCOMES:
The correlation between the maximum perfusion index (PI), the time to reach maximum PI during cuff release and the maximal changes in stroke volume index, cardiac index and perfusion index observed during PLR. | During RIC procedure, as well as during PLR.
  In this context, PI is measured on the arm where the blood pressure cuff is placed. Upon cuff release, both the maximum PI and the time to reach this maximum are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrius Pranskunas, PhD, prof., Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- The Hospital of Lithuanian University of Health Sciences Kauno klinikos, department of Intensive care, Kaunas, Lithuania